CLINICAL TRIAL: NCT00284310
Title: Follow-up of Patients After 4-row Arthrodesis or Proximal Row Carpectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005/183
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2014-12

CONDITIONS: Wrist Surgery
Keywords: Wrist surgery: 4-corner arthrodesis or proximal row carpectomy
MeSH Terms: interventions — Immunologic Memory; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- wrist surgery (Experimental)
  Interventions: Procedure: Anamnesis and clinical examination

INTERVENTIONS:
Procedure: Anamnesis and clinical examination — Anamnesis and clinical examination to follow.

SUMMARY:
The purpose of this trial is to follow-up on patients who underwent different types of wrist surgery: 4-row arthrodesis or proximal row carpectomy.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent wrist surgery (4-row arthrodesis or proximal row carpectomy) between 1998 and 2004

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Results of both types of wrist surgery | 5 to 10 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be